CLINICAL TRIAL: NCT06048588
Title: A Phase I/IIa Trial to Evaluate the Safety, Tolerability, PK, and Preliminary Efficacy of Single and Multiple Ascending Doses of YN001 in Healthy Subjects and Multiple Ascending Doses of YN001 in Patient With Coronary Atherosclerosis
Brief Title: YN001 in Healthy Subjects and Patients With Coronary Atherosclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Inno Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YN001-002
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- YN001 (Experimental): YN001 will be administrated intravenous by single ascending dose, multiple ascending doses weekly or twice a week.
  Interventions: Drug: YN001
- Part I-Matching placebo for YN001 (Placebo Comparator): Matching placebo for YN001 will be administrated intravenous.
  Interventions: Drug: Placebo for YN001
- Part II-Rosuvastatin calcium tablets (Active Comparator): Rosuvastatin calcium tablets will be given by orally.
  Interventions: Drug: rosuvastatin calcium tablets

INTERVENTIONS:
Drug: YN001 — In single ascending dose (SAD) part of study in health subjects, YN001 will be administrated one time with dosage from 10 mg to 120 mg (planned). In multiple ascending doses (MAD) part of study in health subjects, YN001 will be given twice a week from 5 mg to 40 mg up to 15 days. In MAD part of study in patients with coronary atherosclerosis, YN001 will be injected weekly or twice a week from 5mg to 40mg up to 85 days.
  Arms: YN001
Drug: Placebo for YN001 — The injection solution to mimic the YN001
  Other Names: Placebo
  Arms: Part I-Matching placebo for YN001
Drug: rosuvastatin calcium tablets — In MAD part of study in patients with coronary atherosclerosis, Rosuvastatin calcium tablets will be taken orally by 10 mg daily up to 85 days
  Other Names: Crestor®
  Arms: Part II-Rosuvastatin calcium tablets

SUMMARY:
This study consists of two parts. The SAD and MAD of part I are a randomized, double-blind, placebo-controlled, single and multiple ascending dose study in healthy adult subjects. The MAD expansion cohort of part I is single arm and multipal ascending dose in heallthy subjects. Part II (phase Ib/IIa) is a multicenter, randomized, controlled, open label, multiple ascending dose study in patients with coronary atherosclerosis.

DETAILED DESCRIPTION:
Part I (phase Ia) is consists of 2 sections. The sections 1 is designed to evaluate the safety, tolerability, and pharmacokinetics of single and multiple ascending doses of intravenously administered YN001, and to evaluate the effect of SAD of intravenously administered YN001 on the QT/QTc interval, and the immunogenicity of MAD of intravenously administered YN001 in healthy subjects. Besides, the section 2 is designed to evaluate the safety and tolerability of multiple intravenous administration of YN001 without pre-medication or with different pre-medication regimens in Chinese healthy subjects.

Part II (phase Ib/IIa) is designed to evaluate the safety, tolerability, pharmacokinetics, preliminary efficacy, immunogenicity, and the effect on cytokine changes of MAD of intravenously administered YN001 in patients with coronary atherosclerosis.

ELIGIBILITY:
Part I (Phase Ia)-Inclusion criteria:

1. Fully understand the purposes, features, and methods of the study and the possible adverse reactions, voluntarily participate in the study as a subject, and sign the ICF before performing any assessment.
2. Chinese healthy male or female subjects between 18 and 55 years.
3. A Body Mass Index (BMI) of 18-28 kg/m2 (inclusive), with a body weight of at least 50 kg for males and 45 kg for females.
4. Be in good general health at discretion of the investigator based on the results (be normal or abnormal without clinical significance) of medical history, physical examination, vital signs,12-lead ECG, laboratory tests (Hematology; Blood chemistry; Urinalysis, Coagulation and CRP) and viral serology.
5. Female subjects must be non-pregnant and non-lactating, and women of childbearing potential (including the male subject's female companion) must agree to use effective method of contraception from the screening period to 3 months after receiving their last dose of the investigational drug.
6. Willing and able to comply with the requirements of protocol.

Part I (Phase Ia)-Exclusion criteria:

1. Prior treatment with other investigational drug(s) within 3 months or 5 half-lives, whichever is longer, prior to the first dosing.
2. Prior treatment with any prescription drugs, herbal supplements, over the counter (OTC) medication, dietary supplements (vitamins included), or any type of vaccination within 2 weeks prior to the first dosing.
3. Presenting with history of severe food allergy (e.g., anaphylactic reaction). Mild (e.g., non-anaphylactic, hypersensitivity) food allergies such as lactose intolerance/ glucose intolerance are permitted.
4. Allergy to multiple kinds of drugs or presenting with history of allergic reactions to any components of the study drug.
5. Known any clinically abnormal diseases or factors, including but not limited to neurological, cardiovascular, hematological, hepatic, renal, gastrointestinal, respiratory, metabolic, endocrine, immunological, skeletal system diseases, or other reasons that, in the opinion of the investigator, makes the subject inappropriate for inclusion in this study.
6. Presenting with history of myopathy/ myalgia, or susceptible to myopathy/ rhabdomyolysis.
7. Presence of hypothyroidism.
8. Presenting and/or relapse history (within the last 3 years) of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated, or not treated) or cardiac dysfunction or myocardial infarction.
9. Known inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding within 6 months prior to the first dosing.
10. Presenting with history of pancreatic injury or pancreatitis within 6 months prior to the first dosing.
11. Presence of symptoms of urinary obstruction or difficulty in voiding.
12. Presenting and/ or relapse history (within the last 3 years) of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).
13. Evidence of major diseases that not recovered within 2 weeks prior to the first dosing, or major surgery is expected during the study.
14. Presenting with history of impaired renal function defined by clinically significantly abnormal creatinine or BUN and/ or urea values, or abnormal urinary constituents (e.g., albuminuria).
15. Presence of liver disease or liver injury, defined by abnormal liver function tests.
16. Fasting triglyceride > 3.4 mmol/L.
17. Presenting with history of clinically significant ECG abnormalities, or any of the following abnormalities at screening or baseline. QTcF>470 msec for male, QTcF>480 msec for female.
18. Hemoglobin levels are below 120 g/L for males and 110 g/L for females at screening.
19. Donation or blood loss is more than 400 mL within 3 months prior to screening.
20. Use more than 10 cigarettes per day or habitual use of nicotine-containing products within 3 months prior to screening.
21. Presenting with history of drug abuse within 12 months prior to screening, or use of any drugs within 3 months prior to screening, or a positive result of drug abuse screen at screening.
22. Consumption of more than 14 standard drinks of alcohol per week within 3 months prior to screening, or consumption of alcohol-containing products 48 hours prior to the first dosing or having positive alcohol breath test at baseline.
23. Positive for HBsAg, HCV, HIV, TP-Ab.
24. Presence of any other diseases or conditions that, in the opinion of the investigator, would make it unsuitable for the subject to participate in this study.

Part II (Phase Ib/IIa)-Inclusion criteria:

1. Fully understand the purposes, features, and methods of the study and the possible adverse reactions, voluntarily participate in the study as a subject, and sign the ICF before performing any assessment.
2. Chinese male or female subjects between 18 and 75 years.
3. Patients diagnosed with confirmed coronary atherosclerosis and 25-75% stenosis determined by coronary angiography.
4. Suspicion of vulnerable plaque based on clinical practice and determined by OCT examination.
5. Measurable targeted segment by estimation must be at least 40 mm in length.
6. Female subjects must be non-pregnant and non-lactating, and women of childbearing potential (including the male subject's female companion) must agree to use effective method of contraception from the screening period to 3 months after receiving their last dose of the investigational drug.
7. Willing and able to comply with the requirements of protocol.

Part II (Phase Ib/IIa)-Exclusion criteria:

1. Prior treatment with other investigational drug(s) within 30 days or 5 half-lives, whichever is longer, prior to the first dosing.
2. Any type of vaccination within 4 weeks prior to the first dosing.
3. Presence of moderate or heavily calcification lesion in target segment determined by coronary angiography.
4. Known familial hypercholesterolemia.
5. Relapse and highly symptomatic arrhythmia uncontrolled by drugs within the past 3 months, such as ventricular tachycardia, atrial fibrillation with rapid ventricular rate and paroxysmal supraventricular tachycardia.
6. Presenting with history of any type of stroke (cerebral lacunar infarction excluded).
7. Presenting with history of myopathy/ myalgia, or susceptible to myopathy/ rhabdomyolysis.
8. Known inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding within 6 months prior to the first dosing.
9. Presenting with history of pancreatic injury or pancreatitis within 6 months prior to the first dosing.
10. Evidence of major diseases that not recovered within 2 weeks prior to the first dosing, or major surgery is expected during the study.
11. Any surgical operation is planned during the study.
12. Presenting with history of malignancy.
13. Presence of any type of autoimmune disease.
14. Allergy to multiple food or drugs or presenting with history of allergic reactions to any components of the study drug.
15. Prior treatment with CABG, PCI, heart transplantation, SAVR/TAVR, etc., or CABG, PCI, heart transplantation, SAVR/TAVR, etc., is planned during the study.
16. Life expectancy is less than 1 year.
17. Left ventricular ejection fraction (LVEF) <40%.
18. Left main coronary artery disease, defined as left main coronary artery stenosis≥50% by angiographic estimation.
19. Uncontrolled hypertension.
20. Active liver disease or hepatic dysfunction defined by any of ALT, AST, or serum bilirubin exceeding 1.5ULN.
21. Presence of renal insufficiency (eGFR < 30 mL/min/1.73m2).
22. Presence of hypothyroidism.
23. Type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus.
24. Positive for HBsAg, HCV, HIV, TP-Ab.
25. Presence of any other diseases or conditions that, in the opinion of the investigator, would make it unsuitable for the subject to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2025-04-27 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Part I: The safety and tolerability of YN001 in healthy subjects. | Up to 29 days
  To evaluate the incidence of Adverse Events as Assessed by CTCAE v5.0, Clinically Significant Laboratory Abnormalities, Clinically Significant Electrocardiogram Abnormalities, Clinically Significant Vital Signs Abnormalities, Clinically Significant Physical Examination Abnormalities.
Part I: Maximum plasma concentration(Cmax) of YN001 | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects
Part I: Time of maximum concentration (Tmax) of YN001 | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Part I: Elimination half-life (t1/2) of YN001 | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Part I: Area under the plasma concentration-time curve from time 0 to the collection time point of the last measurable concentration (AUC0-t) of YN001 | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Part II: The safety and tolerability of intravenously administered YN001 in patients with coronary atherosclerosis. | Up to 29 days
  To evaluate the incidence of Adverse Events as Assessed by CTCAE v5.0, Clinically Significant Laboratory Abnormalities, Clinically Significant Electrocardiogram Abnormalities, Clinically Significant Vital Signs Abnormalities, Clinically Significant Physical Examination Abnormalities, Clinically Significant Echocardiogram Abnormalities.

SECONDARY OUTCOMES:
Part I: C-QTc analysis | Pre-dose and up to 48 hours post initiation of infusion
  To evaluate the effect of SAD of YN001 on QT/QTc interval prolongation and relationship between YN001 exposure and QT/QTc Interval changes in Chinese healthy subjects.
Part I: Immunogenicity analysis | Up to 96 hours of post initiation of last dose
  To evaluate the immunogenicity of MAD of intravenously administered YN001 in Chinese healthy subjects.
Part I: Pharmacodynamic evaluation | Up to 96 hours of post initiation of last dose
  To evaluate the change LDL-C, HDL-C,TC and TG from baseline to EOT
Part II: Maximum plasma concentration(Cmax) of YN001 | Up to 96 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in patients with coronary atherosclerosis.
Part II: Time of maximum concentration (Tmax) of YN001 | Up to 96 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in patients with coronary atherosclerosis.
Part II: Elimination half-life (t1/2) of YN001 | Up to 96 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in patients with coronary atherosclerosis.
Part II: Area under the plasma concentration-time curve from time 0 to the collection time point of the last measurable concentration (AUC0-t) of YN001 | Up to 96 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in patients with coronary atherosclerosis.
Part II: Change in percent atheroma volume (PAV) of coronary plaque comparing to baseline | Up to 91 days or EOT
  PAV will be determined by intravascular ultrasound (IVUS)
Part II: Change in total atheroma volume (TAV) of coronary plaque comparing to baseline | Up to 91 days or EOT
  TAV will be determined by intravascular ultrasound (IVUS)
Part II: Change in coronary minimal lumen area (MLA) comparing to baseline | Up to 91 days or EOT
  MLA will be determined by intravascular ultrasound (IVUS)
Part II: Change in maximum lipid arc and lipid core length of coronary plaque comparing to baseline | Up to 91 days or EOT
  lipid arc and lipid core length will be determined by optical coherence tomography (OCT)
Part II: Change in minimum fibrous cap thickness (FCT) of coronary plaque comparing to baseline | Up to 91 days or EOT
  FCT will be determined by optical coherence tomography (OCT)
Part II: Change in detection rate of macrophage cluster within coronary plaque comparing to baseline | Up to 91 days or EOT
  detection rate of macrophage cluster will be determined by optical coherence tomography (OCT)
Part II: Change in maximum IMT and plaque thickness | Up to 91 days or EOT
  IMT will be determined by carotid ultrasound scans
Part II: Change in atherosclerosis plaque located at other arteries | Up to 91 days or EOT
  Other arteries plaque will be determined by CTA or MRA
Part II: Immunogenicity analysis | Up to 91 days or EOT
  To evaluate the immunogenicity of MAD of intravenously administered YN001 in Chinese patients with coronary atherosclerosis.
Part II: Cytokines analysis | Up to 91 days or EOT
  To evaluate the effect of MAD of intravenously administered YN001 on Cytokines levels in Chinese patients with coronary atherosclerosis.
Part II： Pharmacodynamic analysis | Up to 91 days or EOT
  Change in LDL-C,HDL-C,TC and TG levels form baseline to EOT

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Chen, Master, Study Director — Beijing Inno Medicine Co., Ltd.
Locations (6):
- China (6):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University first hospital, Beijing, Beijing Municipality
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - First Hospital of Jilin University, Changchun, Jilin
  - Renji Hospital Shanghai Jiaotong Unv. school of Medicine, Shanghai, Shanghai Municipality